CLINICAL TRIAL: NCT05815849
Title: Effect of Enteral Olive Oil Supplement On Weight Gain, Length of Hospital Stay, And Development of Some Complications in Very Low Birth-Weight Infants: A Randomized Controlled Study
Brief Title: Effect of Enteral Olive Oil Supplement On Weight Gain and Development of Some Complications in Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sinem Yalnızoglu Caka, Asst. Prof, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YYB22032023
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Olive Oil Adverse Reaction; Nursing Caries; Enteral and Supplement Feeds Adverse Reaction; Preterm
Keywords: olive oil; neonatal intensive unit; Preterm infant
MeSH Terms: conditions — Premature Birth | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding was used in the study. For this purpose, the participants were not specified in which group they belonged to the research. Therefore, a separate informed consent form was prepared for each group. In order to avoid bias in the analysis of the research data, statistician blinding was also applied. While coding the research data, the research groups were coded as A and B, and the statistician was prevented from knowing which letter represented which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil (Active Comparator): In our unit, according to the recommendations to start and increase enteral feeding in preterm infants in the Turkish Neonatal Society feeding group, Total Parenteral Nutrition (TPN) and Minimal Enteral Nutrition (MEN) are started from the first day. If the infant's weight is between 1000-1500 grams, it is increased to feed the infant as 15-20 ml/kg/day (for 1-2 days) and then 30 ml/kg/day every 2-3 hours. If the infant's weight is between 1500-1800 grams, he/she is fed as 20 ml/kg for 1 day and then 30 ml/kg/day, every 3 hours. BM fortification is initiated when feeding reaches 50-100 ml/kg (recommended 80 ml/kg) [21].At this stage (approximately from the seventh day after starting to take 25-30 ml/kg/day orally), 0.5 cc/30 ml of olive oil (a brand easily available in the markets) was added to the milk at each feeding of the infants in the intervention group.
  Interventions: Dietary Supplement: Olive oil
- Recommendations to start enteral feeding (No Intervention): In our unit, according to the recommendations to start and increase enteral feeding in preterm infants in the Turkish Neonatal Society feeding group, Total Parenteral Nutrition (TPN) and Minimal Enteral Nutrition (MEN) are started from the first day. If the infant's weight is between 1000-1500 grams, it is increased to feed the infant as 15-20 ml/kg/day (for 1-2 days) and then 30 ml/kg/day every 2-3 hours. If the infant's weight is between 1500-1800 grams, he/she is fed as 20 ml/kg for 1 day and then 30 ml/kg/day, every 3 hours. BM fortification is initiated when feeding reaches 50-100 ml/kg (recommended 80 ml/kg) [21].

INTERVENTIONS:
Dietary Supplement: Olive oil — 0.5 cc/30 ml of olive oil (a brand easily available in the markets) was added to the milk at each feeding of the infants in the intervention group
  Arms: Olive oil

SUMMARY:
Objective: The objective of the present research is to compare the nutritional status, weight gain, length of hospital stay, and development of some complications in very low birth-weight (VLBW) infants who received and did not receive olive oil supplementation enterally.

DETAILED DESCRIPTION:
It is known that nutrition of very low birth-weight (VLBW, <1500 g) neonates is as crucial as the treatments they receive in the neonatal intensive care unit to prevent problems that may develop in long-term follow-ups and increase their quality of life. VLBW neonates need parenteral nutrition as an energy source to ensure optimal growth, and lipid emulsion represents an indispensable part of total parenteral nutrition [1]. VLBW neonates with an underdeveloped immune system and antioxidant defense due to preterm birth are vulnerable to oxidative stress, which takes an important part in the development of diseases, e.g., chronic lung disease (CLD), retinopathy of prematurity (ROP), necrotizing enterocolitis (NEC), and intraventricular hemorrhage, which may increase the risk of morbidity [2,3]. Prematurity also causes the insufficient supply of long-chain polyunsaturated fatty acids (LC-PUFAs), including eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), most of which are transferred to the fetus during the third trimester of pregnancy [4]. These LC-PUFAs are essential and important for visual and cognitive development and reducing thrombotic and inflammatory responses [5].

The continuation of intrauterine growth and development in the extrauterine period without interruption may be possible by providing parenteral and enteral nutrition support in the early period and maintaining this support uninterruptedly [6]. Studies have proved that breast milk is the gold standard for feeding neonates under all conditions. However, despite its enormous benefits, unsupplemented breast milk can be nutritionally inadequate for preterm infants for various reasons. First, breast milk does not have a sufficient amount of some nutrients required to ensure the rapid growth of preterm infants [7], and nutrient concentrations can fluctuate over time. Of these, fat is one of the most variable nutrients [8]. Studies have demonstrated that there are temporal and interindividual differences according to the mother's diet, time of day, and breastfeeding duration (e.g., a richer fat content of hindmilk) [9,10]. When breast milk alone cannot meet these needs, it is recommended that special nutritional supplements in the form of powder or liquid be added to breast milk and given to the infant [11].

Due to its content, olive oil has antioxidant, cell regenerative, and anti-carcinogenic properties that help digestion [12]. There are clear pieces of evidence indicating that parenterally administered oil emulsions can be well tolerated by VLBW and even extremely low birth-weight infants from the first day and even from the first 1-2 hours of life [13-15]. The objective of the current research was to compare the nutritional status, weight gain, length of hospital stay, and the development of some complications (BPD, ROP, GIS intolerance, etc.) in preterm neonates who received and did not receive olive oil enterally for calorie support.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants;

* Between the 28th-36th weeks of gestation
* Weighing over 1000 g during the study
* Stable vital signs
* Being able to consume 75% of the total protein and energy through an orogastric tube
* Fed with breast milk and breast milk fortifiers

Exclusion Criteria:

Presence of;

* Necrotizing enterocolitis
* Pneumothorax
* Skull fracture
* Major congenital anomalies
* Suspected or diagnosis of metabolic disease
* History of pathological jaundice (jaundice developing in the first 24 hours),
* History of surgery that might affect the residual
* Using muscle relaxants, analgesics, sedative or inotropic drugs

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
weight gain of preterm infants | up to 6 months
  The infants' weight gain were monitored daily until discharge
length of hospital stay of preterm infants | up to 6 months
  The hospital stays of the control and experimental groups were recorded.
developing prematurity-related complications (Bronkopulmoner displazi (BPD), Retinopathy of prematurity (ROP), Gastric intolerance (GI)) | up to 6 months
  Gastric intolerance (GI) was considered as the inability to digest more than 50% of the enteral nutrition presented as the Gastric Residual Volume (GRV), or abdominal distention and vomiting, or both, and accordingly, the patient's nutritional plan being disrupted [6]. In the findings of ROP, the ROP Diagnosis and Treatment Guidelines were considered, and it was evaluated as severe ROP in case of ROP being stage 3 or higher in both eyes or in case of the infant being treated with laser or antivascular endothelial growth factor therapy [19]. BPD was graded according to the BPD Prevention and Follow-up Guidelines, and all mild/moderate/severe cases were enrolled in the research. Jaundice levels of preterm infants were studied by examining direct bilirubin in the blood. Infants with a history of pathological jaundice were not included in the research [20].

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uauy R, Hoffman DR, Peirano P, Birch DG, Birch EE. Essential fatty acids in visual and brain development. Lipids. 2001 Sep;36(9):885-95. doi: 10.1007/s11745-001-0798-1. PMID 11724460
- [Background] Sharda B. Free radicals: emerging challenge in environmental health research in childhood and neonatal disorders. Int J Environ Res Public Health. 2006 Sep;3(3):286-91. doi: 10.3390/ijerph2006030035. PMID 16968976
- [Background] Lembo C, Buonocore G, Perrone S. Oxidative Stress in Preterm Newborns. Antioxidants (Basel). 2021 Oct 23;10(11):1672. doi: 10.3390/antiox10111672. PMID 34829543
- [Background] Robinson DT, Martin CR. Fatty acid requirements for the preterm infant. Semin Fetal Neonatal Med. 2017 Feb;22(1):8-14. doi: 10.1016/j.siny.2016.08.009. Epub 2016 Sep 3. PMID 27599697
- [Background] Grimm H, Mertes N, Goeters C, Schlotzer E, Mayer K, Grimminger F, Furst P. Improved fatty acid and leukotriene pattern with a novel lipid emulsion in surgical patients. Eur J Nutr. 2006 Feb;45(1):55-60. doi: 10.1007/s00394-005-0573-8. Epub 2005 Jul 22. PMID 16041475
- [Background] Moore TA, Wilson ME. Feeding intolerance: a concept analysis. Adv Neonatal Care. 2011 Jun;11(3):149-54. doi: 10.1097/ANC.0b013e31821ba28e. PMID 21730906
- [Background] Su BH. Optimizing nutrition in preterm infants. Pediatr Neonatol. 2014 Feb;55(1):5-13. doi: 10.1016/j.pedneo.2013.07.003. Epub 2013 Sep 16. PMID 24050843
- [Background] Patel P, Bhatia J. Human milk: the preferred first food for premature infants. Journal of Human Nutrition & Food Science. 2016;4(5):1098.
- [Background] Bhatia J. Human Milk for Preterm Infants and Fortification. Nestle Nutr Inst Workshop Ser. 2016;86:109-19. doi: 10.1159/000442730. Epub 2016 Jun 27. PMID 27347886
- [Background] Amissah EA, Brown J, Harding JE. Fat supplementation of human milk for promoting growth in preterm infants. Cochrane Database Syst Rev. 2020 Aug 25;8(8):CD000341. doi: 10.1002/14651858.CD000341.pub3. PMID 32842164
- [Background] Underwood MA. Human milk for the premature infant. Pediatr Clin North Am. 2013 Feb;60(1):189-207. doi: 10.1016/j.pcl.2012.09.008. Epub 2012 Oct 18. PMID 23178065
- [Background] Lucas L, Russell A, Keast R. Molecular mechanisms of inflammation. Anti-inflammatory benefits of virgin olive oil and the phenolic compound oleocanthal. Curr Pharm Des. 2011;17(8):754-68. doi: 10.2174/138161211795428911. PMID 21443487
- [Background] Thureen PJ. Early aggressive nutrition in very preterm infants. Nestle Nutr Workshop Ser Pediatr Program. 2007;59:193-204; discussion 204-8. doi: 10.1159/000098536. PMID 17245100
- [Background] Drenckpohl D, McConnell C, Gaffney S, Niehaus M, Macwan KS. Randomized trial of very low birth weight infants receiving higher rates of infusion of intravenous fat emulsions during the first week of life. Pediatrics. 2008 Oct;122(4):743-51. doi: 10.1542/peds.2007-2282. PMID 18829797
- [Background] Salama GS, Kaabneh MA, Almasaeed MN, Alquran MIa. Intravenous lipids for preterm infants: a review. Clin Med Insights Pediatr. 2015 Feb 9;9:25-36. doi: 10.4137/CMPed.S21161. eCollection 2015. PMID 25698888
- [Background] Amini E, Shariat M, Nayeri F, et al. A randomized controlled clinical trial of olive oil added to human breast milk for weight gaining in very low birth weight infants. J Family Reprod Health. 2011; 5(3):73-78.
- [Background] Kanik EA, Taşdelen B, Erdoğan S. Klinik Denemelerde Randomizasyon. Marmara Medical Journal. 2011;24(3), 149-155.
- [Background] Satar M, Arisoy AE, Celik IH. Turkish Neonatal Society guideline on neonatal infections-diagnosis and treatment. Turk Pediatri Ars. 2018 Dec 25;53(Suppl 1):S88-S100. doi: 10.5152/TurkPediatriArs.2018.01809. eCollection 2018. PMID 31236022
- [Background] Derneği TN, Derneği TO. Türkiye Prematüre Retinopatisi Rehberi 2021 Güncellemesi. [cited 2022 Aug 27]. Available from: http://www.neonatology.org.tr/wp-content/uploads/2021/08/Turkiye-Premature-Retinopa-tisi-2021-Guncellemesi-1.pdf
- [Background] Derneği TN. Yenidoğan Sarılıklarında Yaklaşım, İzlem ve Tedavi Rehberi 2022 Güncellemesi. [cited 2022 Aug 27]. Available from: http://www.neonatology.org.tr/wp-content/uploads/2022/09/Turk-Neonatoloji-Dernegi-Sarilik-Rehberi-2022-Guncellemesi.pdf
- [Background] Kültürsay N, Bilgen H, Türkyılmaz C. Türk Neonatoloji Derneği Prematüre ve Hasta Term Bebeğin Beslenmesi Rehberi 2018 Güncellemesi. Ankara, Türk Neonatoloji Derneği. [cited 2022 Aug 27]. Available from: https://www.neonatology.org.tr/wp-content/uploads/2020/04/premature_rehber_2018.pdf